CLINICAL TRIAL: NCT04428190
Title: Prebiotic Therapy to Improve Outcomes of Renal Transplant
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The W. Garfield Weston Foundation (Unknown); St. Joseph's Health Care London (Other); London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRT01
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Kidney Transplant; Complications
Keywords: kidney; kidney transplant; prebiotic; human milk oligosaccharide; HMO; renal transplant
MeSH Terms: interventions — Prebiotics; Health Maintenance Organizations

STUDY DESIGN:
Intervention Model Description: One placebo arm and one active treatment arm, participants will be assigned to each arm equally.
Who Masked: Participant, Investigator
Masking Description: No other parties will be masked for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Milk Oligosaccharide (HMO) (Active Comparator): 10 g sachet, self-administered for 3 months.
  2'-O-fucosyllactose and lacto-N-neotetraose, novel human milk oligosaccharide (HMO) sugars have been shown to stimulate the production of short chain fatty acids, especially propionate. Propionate has been shown to be important in attenuating hypertrophy, fibrosis, vascular dysfunction and hypertension (Bartolomaeus H et al 2019Mar12) and extremely important for the gut kidney axis (Li L et al 2017Dec11).
  Interventions: Dietary Supplement: Human Milk Oligosaccharides (HMO)
- Placebo (Placebo Comparator): 10 g sachet, self-administered for 3 months.
  Placebo sachets are identical to the HMO sachets in color, taste, smell, size and shape
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Human Milk Oligosaccharides (HMO) — Sachet containing 10 grams of HMO
  Other Names: Prebiotic
  Arms: Human Milk Oligosaccharide (HMO)
Other: Placebo — Sachet manufactured to mimic 10g of HMO
  Other Names: Placebo for HMO
  Arms: Placebo

SUMMARY:
An investigator initiated pilot study: two arm, double blind, placebo controlled, randomized, group of approximately 60 patients undergoing a kidney transplant. Participants will be treated with human milk oligosaccharide (HMO) prebiotic versus placebo over 12 weeks from start of the investigational medication date (approximately 3 months) to test whether HMO can improve renal transplant outcomes. Participants will be followed up for 3 months after after they complete the treatment portion of the study. HMO sachets will be administered to determine the safety and efficacy of HMO relative to placebo in improving renal transplant outcomes in patients by reducing delayed graft function and side effects from post transplant therapy.

DETAILED DESCRIPTION:
Nearly three million people worldwide suffer from end stage renal disease (ESRD), which has debilitating consequences on the quality of life of patients There is a discrepancy between the availability of organs and the increasing number of patients placed on the waiting list. Canadians with ESRD requiring kidney transplantation has increased by 38% from 2005-2014, whereas the number of transplantable organs has not met this growing need.

As clinicians use more marginal donors, the effects of ischemic injury from the procurement process become more pronounced. This ischemia reperfusion injury (IRI) has been linked to increased delayed graft function, rejection and decreased long-term function. Approximately 20% of transplanted patients subsequently return to dialysis due to poor graft function. Therefore, one of the major goals of the transplant community has now shifted to ensuring the longevity of transplanted organs. Research priorities need to shift towards developing ways to ensure the longevity of grafts through modification of recipient factors.

Patients are also required to remain on immunosuppressive drugs following transplant in order to maintain the graft. These have a variety of side effects, including diarrhea and intestinal malabsorption, which can lead to a lack of patient compliance with post transplant therapy and a reduced quality of life.

Patients with ESRD also have an expansion of bacteria that produce urease and uric acid and produce fewer short-chained fatty acids and vitamins.

This is important as it is theorized that the production of short-chained fatty acids by microorganisms in the GI tract are crucial as both the energy source, and to the maintenance of intestinal permeability, which contribute to a healthy gastrointestinal tract.

The expansion of bacteria that produce urease and uric acid contribute to toxicity and inflammation in the GI tract that can cause complications in these patients.

In order to reduce both delayed graft function and side effects from post transplant therapy, novel support options are required. One option is the use of prebiotics.

Non-digestible sugar prebiotics have potential for use in these patients. The Principal Investigator/Sponsor will test this potential in a pilot clinical study with a Human milk oligosaccharides (HMO) prebiotic mix that have been shown to stimulate the production of short chain fatty acids, especially propionate. Propionate has been shown to be important in attenuating hypertrophy, fibrosis, vascular dysfunction and hypertension and is extremely important for the gut kidney axis. Prebiotics offer a safe and well-tolerated therapy, which could have a positive impact by improving systemic inflammatory responses, improving gut barrier function, helping to reduce immunosuppressive drug side effects and stabilizing its dosing.

This study will assess blood, and urine samples collected as part of the participant's post-transplant follow up at eight time points to determine graft function.

Urine and a faecal sample will be collected at 6 time points for microbiome analyses at baseline, day 7, 30, 60, 120 and 180 from the date of starting the study product. Prior to commencing their treatment, and at days 60,90,150, and 180, the research coordinator (blinded to the randomisation) will assess patients using the SF-36 and GI Health questionnaires during clinic visits, or by telephone interview.

Protocol compliance will be tested through product count and interviews at each follow-up visit. Side effects will be assessed using standardized case report forms at each visit. Participants will be encouraged to report any events they may experience directly to the coordinator.

Participants who withdraw consent to continue treatments, will be encouraged to undergo the planned assessments. Withdrawal at the request of investigators or medical personnel may include, but are not limited to:

1. Symptoms are deemed to be potentially related to the study product
2. New diagnosis of exclusion criteria;
3. Unacceptable side effects;
4. Death

Estimated time to complete recruitment: Averaging 86 weeks, approximately 20 months

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over receiving a kidney transplant.

Exclusion Criteria:

* Under 18 years of age
* Inability to give consent
* Usage of probiotics or other prebiotics.
* Have had carcinomas during the last 5 years
* Bowel surgery
* Crohn ́s disease and other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Short Form Health Survey (SF-36) | 24 weeks
  The Short Form Health Survey will measure participant satisfaction using a scale from 1 - 5, 1 being the best outcome, and 5 being the worst outcome.
Adverse Events | 24 weeks
  Adverse events will be recorded through case report forms and reported to the principal investigator. Side effects will be assessed using standardized case report forms at each visit. Participants are encouraged to contact the coordinator to report any concerns.

SECONDARY OUTCOMES:
Microbiome changes from baseline to end of treatment | 12 weeks
  Changes in the entire bacterial community from baseline to end of study will be assessed in the lab from faecal and urine samples collected by the participant. The microbes may vary by participant and the study will be looking at which ones present themselves in each case. Units of measure via culture are colony forming units per g (cfu/g).
Microbiome changes post intervention | 12 weeks
  Changes in the entire bacterial community after study intervention will be assessed in the lab from faecal and urine samples collected by the participant. The microbes may vary by participant and this outcome measure will be looking at which ones present themselves in each case.

OTHER OUTCOMES:
Number of participants who experience kidney rejection | 24 weeks
  A kidney rejection will be recorded in the adverse event form for the study.
Immunosuppression suppressive drug dose | post-operative day 1, 7, 30, 60, 90, 120, 150 and 180
  will be assessed by the clinic on post-operative day 1, 7, 30, 60, 90, 120, 150 and 180
Infectious complications | post-operative day 30, 60, 90, 120, 150 and 180.
  Cytomegalovirus will be tested by the clinic, typically reported in IU/mL
Serum creatinine | 24 weeks.
  Will be used to determine graft function, and is reported in μmol/L.
Cystatin-c levels | 24 weeks.
  Will be used to determine graft function, and is reported in mg/l.
Estimated glomerular filtration rate (eGFR) | 24 weeks.
  Will be used to determine graft function, and is reported in mL/min/1.73m**2.
Urine output | 24 weeks.
  Will be used to determine graft function, and is reported in mL/day.
Urine protein/creatinine ratio | 24 weeks.
  Will be used to determine graft function, and is reported in g/L
Dialysis episodes | 24 weeks.
  Will be used to determine graft function, and will be measured by the amount of times a participant required dialysis.
Renal micro-perfusion using Doppler ultrasound | 24 weeks.
  Will be used to determine graft function by providing an assessment of vascular changes.
Search Results Web results Kidney Injury Molecule-1 (Kim-1) | 24 weeks.
  Will be used to determine graft function, and is reported in ng/ml
Neutrophil gelatinase-associated lipocalin (NGAL) | 24 weeks.
  Will be used to determine graft function, and is reported in ng/ml
Immunosuppression drug serum levels (MMF and FK-506) | post-operative day 1, 7, 30, 60, 90, 120, 150 and 180
  will be assessed by the clinic, typically reported in mg/ml.
Serial viral serologies | post-operative day 30, 60, 90, 120, 150 and 180.
  Polyomavirus will be tested by the clinic post-op, typically reported in IU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Alp Sener, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pluznick JL. Gut microbiota in renal physiology: focus on short-chain fatty acids and their receptors. Kidney Int. 2016 Dec;90(6):1191-1198. doi: 10.1016/j.kint.2016.06.033. Epub 2016 Aug 26. PMID 27575555
- [Background] Lee JR, Muthukumar T, Dadhania D, Taur Y, Jenq RR, Toussaint NC, Ling L, Pamer E, Suthanthiran M. Gut microbiota and tacrolimus dosing in kidney transplantation. PLoS One. 2015 Mar 27;10(3):e0122399. doi: 10.1371/journal.pone.0122399. eCollection 2015. PMID 25815766
- [Background] Elison E, Vigsnaes LK, Rindom Krogsgaard L, Rasmussen J, Sorensen N, McConnell B, Hennet T, Sommer MO, Bytzer P. Oral supplementation of healthy adults with 2'-O-fucosyllactose and lacto-N-neotetraose is well tolerated and shifts the intestinal microbiota. Br J Nutr. 2016 Oct;116(8):1356-1368. doi: 10.1017/S0007114516003354. Epub 2016 Oct 10. PMID 27719686
- [Background] Harvie RM, Chisholm AW, Bisanz JE, Burton JP, Herbison P, Schultz K, Schultz M. Long-term irritable bowel syndrome symptom control with reintroduction of selected FODMAPs. World J Gastroenterol. 2017 Jul 7;23(25):4632-4643. doi: 10.3748/wjg.v23.i25.4632. PMID 28740352
- [Background] Dubberke ER, Riddle DJ; AST Infectious Diseases Community of Practice. Clostridium difficile in solid organ transplant recipients. Am J Transplant. 2009 Dec;9 Suppl 4(0 4):S35-40. doi: 10.1111/j.1600-6143.2009.02891.x. PMID 20070693
- [Background] Rayes N, Seehofer D, Theruvath T, Schiller RA, Langrehr JM, Jonas S, Bengmark S, Neuhaus P. Supply of pre- and probiotics reduces bacterial infection rates after liver transplantation--a randomized, double-blind trial. Am J Transplant. 2005 Jan;5(1):125-30. doi: 10.1111/j.1600-6143.2004.00649.x. PMID 15636620
- [Background] Sawas T, Al Halabi S, Hernaez R, Carey WD, Cho WK. Patients Receiving Prebiotics and Probiotics Before Liver Transplantation Develop Fewer Infections Than Controls: A Systematic Review and Meta-Analysis. Clin Gastroenterol Hepatol. 2015 Sep;13(9):1567-74.e3; quiz e143-4. doi: 10.1016/j.cgh.2015.05.027. Epub 2015 Jun 2. PMID 26044318
- [Background] Lobb I, Jiang J, Lian D, Liu W, Haig A, Saha MN, Torregrossa R, Wood ME, Whiteman M, Sener A. Hydrogen Sulfide Protects Renal Grafts Against Prolonged Cold Ischemia-Reperfusion Injury via Specific Mitochondrial Actions. Am J Transplant. 2017 Feb;17(2):341-352. doi: 10.1111/ajt.14080. Epub 2016 Nov 29. PMID 27743487
- [Background] Al KF, Bisanz JE, Gloor GB, Reid G, Burton JP. Evaluation of sampling and storage procedures on preserving the community structure of stool microbiota: A simple at-home toilet-paper collection method. J Microbiol Methods. 2018 Jan;144:117-121. doi: 10.1016/j.mimet.2017.11.014. Epub 2017 Nov 16. PMID 29155236
- [Background] Bao Y, Al KF, Chanyi RM, Whiteside S, Dewar M, Razvi H, Reid G, Burton JP. Questions and challenges associated with studying the microbiome of the urinary tract. Ann Transl Med. 2017 Jan;5(2):33. doi: 10.21037/atm.2016.12.14. PMID 28217698
- [Result] Perico N, Cattaneo D, Sayegh MH, Remuzzi G. Delayed graft function in kidney transplantation. Lancet. 2004 Nov 13-19;364(9447):1814-27. doi: 10.1016/S0140-6736(04)17406-0. PMID 15541456
- [Result] Wong J, Piceno YM, DeSantis TZ, Pahl M, Andersen GL, Vaziri ND. Expansion of urease- and uricase-containing, indole- and p-cresol-forming and contraction of short-chain fatty acid-producing intestinal microbiota in ESRD. Am J Nephrol. 2014;39(3):230-237. doi: 10.1159/000360010. Epub 2014 Mar 8. PMID 24643131
- [Result] Bartolomaeus H, Balogh A, Yakoub M, Homann S, Marko L, Hoges S, Tsvetkov D, Krannich A, Wundersitz S, Avery EG, Haase N, Kraker K, Hering L, Maase M, Kusche-Vihrog K, Grandoch M, Fielitz J, Kempa S, Gollasch M, Zhumadilov Z, Kozhakhmetov S, Kushugulova A, Eckardt KU, Dechend R, Rump LC, Forslund SK, Muller DN, Stegbauer J, Wilck N. Short-Chain Fatty Acid Propionate Protects From Hypertensive Cardiovascular Damage. Circulation. 2019 Mar 12;139(11):1407-1421. doi: 10.1161/CIRCULATIONAHA.118.036652. PMID 30586752
- [Result] Li L, Ma L, Fu P. Gut microbiota-derived short-chain fatty acids and kidney diseases. Drug Des Devel Ther. 2017 Dec 11;11:3531-3542. doi: 10.2147/DDDT.S150825. eCollection 2017. PMID 29270002
- [Derived] Cooper TE, Scholes-Robertson N, Craig JC, Hawley CM, Howell M, Johnson DW, Teixeira-Pinto A, Jaure A, Wong G. Synbiotics, prebiotics and probiotics for solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 20;9(9):CD014804. doi: 10.1002/14651858.CD014804.pub2. PMID 36126902